CLINICAL TRIAL: NCT03569917
Title: Identification of Gut Microbiome Biomarkers Associated to Acquisition of Enterobacteriae Highly Resistant to Third Generation Cephalosporines Following Ceftriaxone Treatment.
Acronym: ARCMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 143 patients have been recruited instead of 150 but the theoretical date of end of inclusions being reached, we have decided to not prolong again the study.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC17_0462
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Patients Receiving Ceftriaxone in Hospital Emergency Unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient under Ceftriaxone treatment (Experimental)
  Interventions: Other: Rectal swab collection

INTERVENTIONS:
Other: Rectal swab collection — Rectab swab collection will be performed at inclusion and 5 and 30 days later.

SUMMARY:
Patients receiving Ceftriaxone 1 gram or 2 grams per day during their presence in emergency unit of hospital whatever their medical condition, will be included.

Rectal swabs will be collected at inclusion and at days 5 and 30 to perform analysis.

Analysis will be performed to characterize gut microbiome in order to detect intestinal microbiome profiles significantly associated with protection against colonization by third generation cephalosporin resistant Enterobacteriae.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Able to comply with study requirement and to provide informed consent
* Outside the context of tutorship and / or guardianship, affiliated to the Social Security Regime and having consented to participate in the ARCMI study.
* Patient receiving ceftriaxone (1 gram or 2 grams per day) in the emergency department

Exclusion Criteria:

* Patients with acute anorectal pathology incompatible with the swabbing strategy or digital rectal examination.
* Prescription of another dosage of ceftriaxone (more than 2 grams per day)
* Patient with inflammatory bowel disease
* Allergy or contraindication to betalactamines and cephalosporins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Identification of gut microbiome biomarkers | 30 days
  The use of culture-independent techniques, metagenomics and metabolomics, will allow an exhaustive analysis of the intestinal microbiome in order to detect intestinal microbiome profiles (including species, modules, metabolites) significantly associated with protection against colonization by Enterobacteriae resistant to Cephalosporine. Acquisition of a risk index to Enterobacteriae resistance to third generation cephalosporin will be measured by the method developed by Montassier et al, 2016, Genome medicine.

SECONDARY OUTCOMES:
Identification of gut microbiome biomarkers | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes university Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No